CLINICAL TRIAL: NCT02492581
Title: Use of Selincro and Impact on Usual Practice
Acronym: USE-PACT
Status: Completed | Type: Observational
Sponsor: University of Bordeaux (Other)
Collaborators: Lundbeck France (Unknown)
Responsible Party: Principal Investigator, Patrick BLIN, Doctor, University of Bordeaux
Other Study IDs: #16117N
Record Dates: First submitted 2015-07-01; First posted 2015-07-08 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Alcohol Dependence
Keywords: Selincro; cohort; real-life; total alcohol consumption; heavy drinking days; clinical global impression-severity; EQ5D; AQoLS; Sheehan disability scale
MeSH Terms: conditions — Alcoholism | interventions — nalmefene

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Nalmefene — No intervention on the use of Selincro. The physician will prescribe Selincro following its usual practice.
  Other Names: Selincro

SUMMARY:
USE-PACT is a cohort study of patients initiating Selincro® with one-year follow-up, performed using a random sample of prescribers. The aim of the study is to evaluate the use of Selincro in real-life and its impact on alcohol consumption at one year.

DETAILED DESCRIPTION:
Selincro® (nalmefene) has obtained European market authorisation and is indicated "for the reduction of alcohol consumption in adult patients with alcohol dependence who have a high drinking risk level, without physical withdrawal symptoms and who do not require immediate detoxification". The French health authorities (Haute Autorité de Santé, HAS, and Agence Nationale de Sécurité du Médicament et des produits de santé, ANSM) have requested an evaluation of the real-life conditions of use of Selincro and its impact on morbidity.

In response, USE-PACT has been developed : a cohort of patients initiating Selincro® with one-year follow-up.

The primary objective is to evaluate the change of alcohol consumption at one year in patients initiating Selincro® in usual practice.

The secondary objectives are :

* Describe prescriber characteristics,
* Describe the initial demographic, clinical, and biological characteristics of patients at the start of treatment,
* Describe patient support, notably psychosocial, at start of treatment and during treatment,
* Describe characteristics of Selincro® treatment during the study period,
* Describe the frequency of adverse effects during Selincro® treatment.

It is a prospective cohort of patients initiating Selincro® performed using a random sample of general practitioners (GPs), psychiatrists and physicians practicing in specialised structures.

600 patients are required to obtain precision of ± 5 % for the relative variation in alcohol consumption in g/day at one year, with standard deviation of 63% and 95% confidence intervals, i.e. 1000 patients to be included taking into account 40% loss-to-follow-up.

2500 GPs and 2500 psychiatrists will be contacted with the hypothesis of 10% accepting and 7% active physicians and all physicians/specialised structures from the directory of the French alcohology society. It is thus expected 175 GPs, 175 psychiatrists and 85 physicians practicing in specialised structures, based on the hypothesis of an average 2 patients per GP and psychiatrist, and 4 for physicians practicing in specialised structures.

Each participating physician should, during a 4-month period:

* Include in the cohort all patients for whom he/she initiates Selincro® treatment and fulfilling the eligibility criteria, with a maximum of 6 patients per physician;
* Record in a non-inclusion register patients for whom Selincro® is initiated and not included in the cohort, with a maximum of 10 patients per physician;

The physician will do a clinical evaluation at the time of inclusion and will follow the patients included in the cohort according to usual practice, with a clinical evaluation at 1 month ± 8 days (M1), 3 months ± 15 days (M3), 6 months ± 30 days (M6), 9 months ± 30 days (M9), and 12 months ± 30 days (M12) performed during usual follow-up consultations.

In parallel, each included patient will also complete a self-administered questionnaire at the the time of the inclusion. Then, they will receive and complete the self-administered questionnaire at the 5 follow-up periods (M1, M3, M6, M9 and M12).

Patients declared as lost-to-follow-up and, if required, his/her general practitioner will be contacted by telephone by the coordinating centre in order to fill-out a "last known status questionnaire". For patients who could not be reached, vital status will be investigated using the INSEE/INSERM centralised procedure as defined by decree.

A descriptive analysis using SAS® software will be conducted on the basis of a detailed statistical analysis plan developed and submitted for validation to the scientific committee before analysis, according to the following principles:

* For the total population, and in according to prescriber speciality (GP, psychiatrists, physicians practicing in specialised structures), and the existence or not of previous medicinal treatment;
* "Flow chart" presenting the process of physician recruitment and patient inclusion;
* Description of prescriber characteristics;
* Description of treated patients;
* Description of the change in alcohol consumption (primary and secondary criteria):

  * Principal analysis with multiple imputation of missing data for patients followed one year with missing Total Alcohol Consumption (TAC)/Heavy Drinking Days (HDD),
  * First sensitivity analysis without multiple imputation,
  * Second sensitivity analysis with multiple imputation of missing data for patients followed one year with missing TAC/HDD as well as those lost-to-follow-up;
* Description of follow-up;
* Description of Selincro® treatment;
* Description and frequency of adverse events.

Representativeness:

* Comparison of characteristics common to included patients and those in the registry;
* Comparison of initial characteristics of patients followed at 1 year and those not followed at 1 year;
* Comparison of the characteristics of patients included in the cohort with respect to patients extracted from the national health insurance database (EGB: Echantillon Généraliste des Bénéficiaires). Adjustments could be performed if an imbalance with respect to EGB data in order to produce representative data.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years) initiating Selincro
* Patient accepting to participate
* Patient without linguistic barrier, notably to read the information letter and to complete the self-administrated questionnaires
* Patient not included in another study susceptible to modify patient care
* Patient not under a guardianship

Exclusion Criteria:

* Minor patient (≤18 years)
* Patient refusing to participate
* Patient with linguistic barrier
* Patient included in another study susceptible to modify patient care
* Patient under a guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients initiating Selincro because of alcohol dependence
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Relative change of Total Alcohol Consumption (TAC) between inclusion and end of follow-up at one year | One year

SECONDARY OUTCOMES:
Relative and absolute change of TAC with respect to inclusion | at 1 month, 3 months, 6 months, 9 months and 12 months after inclusion
At least 70% reduction in TAC with respect to inclusion | at 1 month, 3 months, 6 months, 9 months and 12 months after inclusion
Change in the alcohol consumption risk level according to the WHO with respect to inclusion | at 1 month, 3 months, 6 months, 9 months and 12 months after inclusion
Relative and absolute change of Heavy Drinking Days (HDD) with respect to inclusion | at 1 month, 3 months, 6 months, 9 months and 12 months after inclusion

OTHER OUTCOMES:
Change in CGI-Severity with respect to inclusion (according to the physician (CGI-S) & according to the Patient (CGI-P)) | at 1 month, 3 months, 6 months, 9 months and 12 months after inclusion
Proportion of patients having attained alcohol consumption objective defined at previous consultation | at 1 month, 3 months, 6 months, 9 months and 12 months after inclusion
Change in family and socio-professional impact (Sheehan Disability Scale) with respect to inclusion | at 1 month, 3 months, 6 months, 9 months and 12 months after inclusion
Change in generic quality of life EQ5D with respect to inclusion | at 1 month, 3 months, 6 months, 9 months and 12 months after inclusion
Change in alcohol quality of life (AQoLS short version with 7 items) with respect to inclusion | at 1 month, 3 months, 6 months, 9 months and 12 months after inclusion
Change in hepatic parameters, collected according to usual practice by the physician with respect to inclusion | at 1 month, 3 months, 6 months, 9 months and 12 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas MOORE, Professor, Study Director — University of Bordeaux
Locations (1):
- University of Bordeaux, Bordeaux, France